CLINICAL TRIAL: NCT01501331
Title: Multiparametric Evaluation of Heart Failure in Device-implanted Patients.
Brief Title: Multiparametric Heart Failure Evaluation in Internal Cardioverter Defibrillators (ICD) Patients
Acronym: MULTITUDE-HF
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giovanni B Forleo, MD, PhD, University of Rome Tor Vergata
Other Study IDs: PTVCARDIO2011_01
Record Dates: First submitted 2011-12-06; First posted 2011-12-29 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Cardiac Resynchronization Therapy; Internal Cardioverter Defibrillators
MeSH Terms: conditions — Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RRT diagnostic tool: Patients implanted with an Energen device or successor.
  Interventions: Device: CRTD or ICD (Energen)

INTERVENTIONS:
Device: CRTD or ICD (Energen) — RRT measurement by cardiac resynchronization therapy devices and implantable cardioverter defibrillators

SUMMARY:
The Boston Scientific Energen family is capable of measuring the respiratory rate trend (RRT) on a daily basis and transmission of data via the Remote Monitoring technology. This may result in early detection of imminent decompensation at a presymptomatic stage. The study will assess the respiratory trends correlation with clinically relevant heart failure events.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for 1-, 2- or 3-chamber ICD implantation according to current guidelines or patient already implanted within the past 45 days with a Energen device or successor
* Able to provide written informed consent

Exclusion Criteria:

* Life expectancy <12 months
* Anticipated non-compliance with the follow-up scheme
* Moderate to severe Chronic Obstructive Pulmonary Disease
* Primary pulmonary hypertension

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients implanted with an Energen device or successor using the RRT diagnostic tool
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Prediction by RRT of cardiovascular death or rehospitalization for worsening of heart failure symptoms. | 24 months
  Respiratory rate changes (maximum, median and minimum values) before a primary event (3-, 2-, 1-week before and on the day of the event) will be compared to those at baseline (6 weeks prior the event).
  Pts with less than 30-day of RR data or events without sufficient baseline will be excluded from the analysis

SECONDARY OUTCOMES:
Proportion of in-hospital consultations with relevant findings (i.e. necessitating changes in medical therapy, device programming or re-hospitalisations/ interventions) | 24 months
  Respiratory rate changes (maximum, median and minimum values) before the event (3-, 2-, 1-week before and on the day of the event) will be compared to those at baseline (6 weeks prior the event).
  Pts with less than 30-day of RR data or events without sufficient baseline will be excluded from the analysis
Correlation of RRT with appropriate ICD therapy (ATP or Shock) | 24 months
  Respiratory rate changes (maximum, median and minimum values) before the event (3-, 2-, 1-week before and on the day of the event) will be compared to those at baseline (6 weeks prior the event).
  Pts with less than 30-day of RR data or events without sufficient baseline will be excluded from the analysis
Correlation of RRT with atrial and ventricular arrhythmias | 24 months
  Respiratory rate changes (maximum, median and minimum values) before the event (3-, 2-, 1-week before and on the day of the event) will be compared to those at baseline (6 weeks prior the event).
  Pts with less than 30-day of RR data or events without sufficient baseline will be excluded from the analysis

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni B Forleo, MD, PhD, Principal Investigator — University of Rome Tor Vergata; Luca Santini, MD, PhD, Principal Investigator — University of Rome Tor Vergata
Locations (2):
- Italy (2):
  - Milan
  - Rome